CLINICAL TRIAL: NCT03122782
Title: Hemostatic Effect of Intrauterine Instillation Of Tranexamic Acid In Hysteroscopic Myomectomy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Hajer Soliman, Resident, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: ASU-2016-2
Record Dates: First submitted 2017-03-06; First posted 2017-04-21 (Actual); Last update posted 2017-06-29 (Actual); Status verified 2017-03

CONDITIONS: Surgical Blood Loss; Fibroid
MeSH Terms: conditions — Blood Loss, Surgical; Leiomyoma | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tranexamic acid (TXA) Group (Active Comparator): Subjects in the Tranexamic acd (TXA) group will receive intrauterine instillation of 500 mg (100mg/ml) Tranexamic acid per 500 ml normal salin (distention medium) during Hysteroscopic Myomectomy.
  Interventions: Drug: Topical application Tranexamic acid
- Normal Saline (control group) (Placebo Comparator): Subjects in the control group will receive 500 ml intrauterine instillation of normal saline with the distention medium (normal saline) during Hysteroscopic Myomectomy.
  Interventions: Drug: Placebo (Normal saline)

INTERVENTIONS:
Drug: Topical application Tranexamic acid — Tranexamic acid (TXA) will be injected to distinction media during hysteroscopy in myomectomy
  Other Names: KAPRON (AMOUN Pharmaceutical co.)
  Arms: Tranexamic acid (TXA) Group
Drug: Placebo (Normal saline) — 5ml of normal saline will be added to every 500 ml of distension media
  Arms: Normal Saline (control group)

SUMMARY:
Study Design:

Randomized Controlled Clinical Trial.

Study Population:

The study population will be a consecutive series of participants attending the Early Cancer Detection Unit (ECDU) at Ain Shams University Maternity Hospital.

80 women who are scheduled to undergo a hysteroscopic myomectomy will be included and will be randomized into two groups:

Group A: women will undergo a hysteroscopic myomectomy with the use of (TXA) Kapron in the distention medium

Group B: women will undergo hysteroscopic myomectomy with the use of placebo(normal saline in the distention medium).

Randomization will be performed using a Computer-generated randomization system.

The allocated groups will be concealed in serially-numbered sealed opaque envelopes that will only be opened after recruitment.

Patient allocation will be performed prior to the induction of anesthesia by an independent person, who will not otherwise be involved in this study.

The trial will be appropriately blinded; the participants, outcome assessors and the surgeon performing the procedure will be blinded to the medication type, which will be used inside the distention medium.

Therefore, this study will be a randomized double blind prospective clinical

Methodology:

1. Informed written consent obtained from the participant.
2. History

   1. Personal history
   2. Menstrual history
   3. Detailed obstetric history
   4. Surgical intervention especially uterine surgeries and any post-operative complication
   5. History of drug intake, especially hormonal treatment or anticoagulant therapy.
3. Routine preoperative investigations in addition to a serum pregnancy test if pregnancy is suspected.
4. Physical examination including general, abdominal and pelvic examination.
5. Hysteroscopy will be performed in the early proliferative phase using normal saline as a distention medium.
6. Only in intervention group (TXA group) KAPRON (Tranexamic acid) will be added to the injected media.

   * In intervention group 500 mg of Kapron for every 500 ml of distending media will be added.
   * In the control group, placebo .i.e. ,normal saline in the same form will be injected inside every 500 ml of the distention medium.
7. The trial will be appropriately blinded; the participants, outcome assessors and the surgeon performing the procedure will be blinded to the medication type, which will be used inside the distention medium. Therefore, our study will be a randomized double blind prospective clinical trial.
8. Intraoperative bleeding and quality of view will be observed.
9. A blood sample will be taken from each participant in both groups after 24 hours from the end of the operation for both hemoglobin and hematocrit levels.

Types of outcome measures:

Primary outcome measures:

Estimated Blood loss defined as comparing the hematocrit and hemoglobin at base line (preoperative ) and 24 hours after surgery with the Tranexamic acid compared to the control group.

Secondary outcome measures:

The quality of view, duration of surgery, the volume of injected media, intraoperative complications and the success of the completion of the operation will be secondary outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be able to understand, and read and sign the study specific informed consent after fully explanation the nature of the study .
2. Subjects exhibit submucous myoma that are completely within the endometrial cavity or extend less than 50 percent into the myometrium (type 0,i)according to European Society Of Hysteroscopy (ESH).
3. The submucous myoma are less than 4 cm in diameter

Exclusion Criteria:

1. Pregnancy
2. Active Pelvic Infection
3. Present or History of Cervical or Uterine Caner
4. Bleeding Diathesis or patient on anticoagulant
5. Contraindication and /or allergy to medication specified in the treatment protocol
6. History of ischemic heart disease
7. Patient with Cardiopulmonary, Hepatic , and renal diseases
8. Patient with metabolic disorders including diabetes
9. Patients with uterine septum or structural abnormality

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-08-01 (Estimated); Primary Completion 2017-08 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Estimated blood loss by comparing changes in hemoglobin level | 24 Hours
  Estimated blood loss by comparing changes in hemoglobin level before hysteroscopic myomectomy (preoperative) and 24 hours after hysteroscopic myomectomy (postoperative) in Tranexamic acid group comparing to the control group
Estimated blood loss by comparing changes in hematocrit level | 24 hours
  Estimated blood loss by comparing changes in hematocrit level before hysteroscopic myomectomy (preoperative) and 24 hours after hysteroscopic myomectomy (postoperative) in the Tranexamic acid group comparing to the control group

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Khairyy Makled, MD, Study Chair — Ain Shams University; Amgad Said Abu-Gamra, MD, Study Chair — Ain Shams University; Radwa Ali Rasheedy, MD, Study Director — Ain Shams University; Hajer Giuma Soliman, M.B.B.CH, Principal Investigator — Ain Shams University